CLINICAL TRIAL: NCT04472325
Title: The Differential Diagnosis and Prognosis of Idiopathic and Atypical Parkinson Disease by Using Diffusion MRI
Status: Completed | Type: Observational
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Wang . Jiun-Jie, Study Principal Investigator, Chang Gung Memorial Hospital
Other Study IDs: 106WFD2650309
Record Dates: First submitted 2020-06-14; First posted 2020-07-15 (Actual); Last update posted 2021-08-06 (Actual); Status verified 2021-08

CONDITIONS: Parkinson Disease
Keywords: Magnetic Resonance Imaging; Neurodegeneration disease; Cognitive impairment; Diagnosis; Prognosis
MeSH Terms: conditions — Parkinson Disease; Cognitive Dysfunction; Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Atypical Parkinson's Disease patients: This group consists of patients includes 35 patients with Progressive Supranuclear Paralysis (PSP), 35 patients with Multiple System Atrophy (MSA), and 35 patients with Cortico-Basal Degeneration (CBD).
- Idiopathic Parkinson's Disease patients: This group consists of patients starting from 2012 to 2013 and includes 87 patients with typical Parkinson's Disease (PD)
- Healthy volunteers: The 96 healthy volunteers should meet the following criteria:
  1. Between 50-80 years old
  2. Right-handed
  3. MMSE score greater than or equal to 26
  4. Able to understand study requirements and give informed consent

SUMMARY:
The hypothesis is that the differential extent of microstructural damages in the affected brain regions can be specific to the disease of interest and could reflect the clinical severity. Therefore, we propose that the whole brain parcellation of diffusion MRI can be used to improve the diagnosis and prediction of clinical outcomes in Parkinson's Disease.

1. A regression model between clinical severity and two-year clinical outcomes and diffusion properties from multiple parcellated regions will be developed.
2. Blind validation will be performed.

DETAILED DESCRIPTION:
Parkinson's disease (PD) is a common progressive neurodegenerative disorder characterized by resting tremor, bradykinesia, restricted mobility, and postural instability. Early diagnosis of PD would be paramount for further treatment and prognosis. The most common neurodegenerative parkinsonian syndrome is known as Parkinson's disease (PD) or idiopathic Parkinson syndrome, if it occurs sporadically (not familial) and its lead clinical symptom is a movement disorder after brainstem-predominant α-synuclein deposition. To distinguish them from Parkinson's disease, other sporadic entities have been named atypical parkinsonian syndromes or atypical parkinsonism. The present review article describes current standards for the diagnosis and treatment of the most important disease entities in this latter group: dementia with Lewy bodies (DLB), multiple system atrophy (MSA), progressive supranuclear palsy (PSP), and corticobasal degeneration (CBD).

PD is diagnosed mainly by neurologists, based on clinical symptoms. However, there are no objective criteria available for their diagnosis. Although magnetic resonance imaging (MRI) is often employed in conjunction with clinical judgment, the images are mostly used to eliminate other diseases, rather than to confirm the diagnosis. Other imaging methods, such as Positron Emission Tomography or Computed Tomography, may help in the diagnosis of PD but have harmful effects on the human body. MRI image of patients with Parkinson's disease is usually normal. Previous studies have also indicated that brain-related areas, such as the atrophy of basal ganglia, are not observed until a period of disease progression. However, the shrinkage of brain tissue cannot be used as a criterion for the diagnosis of Parkinson's disease, because many other diseases are accompanied by atrophy of brain tissue as well. Furthermore, because human brain cells cannot regenerate, It is too late to diagnose or treat when a large number of nerve cells are apoptotic. Since we expect the function of the diseased cells to change first, therefore, if you can detect changes in the patient's brain microenvironment, it is possible to achieve early detection of Parkinson's disease. Magnetic resonance imaging can detect functional images and display functional changes, thus providing an opportunity to detect abnormalities and diagnose diseases early. One of the key technologies in the measurement of functional images is diffusion magnetic resonance imaging.

Diffusion MRI has been widely utilized to investigate the patterns of neural connectivity. Mean diffusivity (MD) and the directionality (fractional anisotropy (FA)) have been studied in epilepsy, multiple sclerosis, and noticeably in Parkinson's Disease. Owing to their paramount pathogenetic role in Parkinson's disease, the basal ganglia in general and the substantia nigra pars compacta, in particular, have been the subject of intense MRI investigation.

The plan uses standard anatomic labeling (AAL) to perform whole-brain diffusion MRI to obtain diffusion data for the whole brain parcellation. We will use statistical methods to identify the areas affected by each PD's subtype, we will also identify areas that are likely to be related to the severity of the disease, and then combine these areas for linear regression analysis. We anticipate that diffusion magnetic resonance imaging can be used as a differential diagnosis, as well as to define areas of high correlation with clinical severity, and to be used for accurate disease prediction and future development, and to provide physicians and patients with clinically important information.

The program uses diffusion magnetic resonance imaging to assess clinical status and prognosis for Parkinson's disease. Our research goal is

1. Establish objective and clear imaging diagnostic criteria of diffusion MRI for idiopathic and atypical Parkinson's disease.
2. Establish objective and clear clinical severity and the prognosis prediction mode of diffusion MRI for idiopathic and atypical Parkinson's disease.

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

* Cardiac pacemaker or defibrillator implantation Intracranial metal device implantation
* Other major systemic diseases, such as renal failure, heart failure, stroke, AMI/unstable angina, poorly controlled diabetes mellitus, poorly controlled hypertension
* Alcohol or drug abuse
* Moderate to severe dementia
* Severe movement disorders
* Imaging data is similar to a nuclear medical examination, exclusion criteria is any abnormality that may affect cognitive function as reflected in computer tomography or MRI records, such as hydrocephalus or encephalitis. Mild cortical atrophy is acceptable.
* History of intracranial surgery including thalamotomy, pallidotomy, and/or deep brain stimulation
* Major physical or neuropsychiatric disorders
* Structural abnormalities that may cause dementia, such as cortical infarction, tumour, or subdural hematoma
* Besides medication for Parkinson's Disease, taking other medication with substances that can pass through the blood-brain barrier
* Besides medication for Parkinson's Disease, taking other medication for more than 10 years
* Treatments or concurrent illnesses other than Alzheimer's Disease that could interfere with cognitive function
* Meet the criteria for dementia (DSM-IV)
* Head trauma with loss of consciousness greater than 10 minutes
* Severe loss of sensation

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All subjects should meet the following criteria:
  1. Between 50-80 years old
  2. Right-handed
  3. Able to understand study requirements and give informed consent
  4. Agree to return for follow-up checks
  5. Able to suspend intake of medication for at least 12 hours
Sampling Method: Non-Probability Sample
Enrollment: 288 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2018-08-01 (Actual); Study Completion 2020-07-31 (Actual)

PRIMARY OUTCOMES:
An objective image-based evidence for the diagnosis, differential diagnosis and prognosis of Parkinson's Disease | end of the third year
  The following will be measured for the diagnostic performance of diffusion MRI:
  1. Regression between cognitive performance and baseline diffusion MRI using Pearson correlation
  2. Leave one out cross validation

SECONDARY OUTCOMES:
prognosis | end of the third year
  To predict the outcome of patient with PD using the diffusion MRI at baseline
prognosis | end of the third year
  Methods for evaluation of worsening cognitive function in neurodegenerative disease
differential diagnosis | end of the second year
  To differentiate patient of PD from PD + using diffusion MRI
Imaging | end of the third year
  High-quality diffusion MRI and image data restoration
Imaging | end of the third year
  High-quality diffusion MRI imaging standards, parcellation methods and image processing protocol

CONTACTS AND LOCATIONS:
Locations (1):
- ChangGung Memorial Hospital, Linkou, Taoyuan District, Taiwan